CLINICAL TRIAL: NCT06067542
Title: Evaluation of the Clinical and Microbiological Effects of Chlorhexidine Toothpaste on Wound Healing Following Tooth Extraction
Brief Title: Effects of Chlorhexidine Toothpaste on Wound Healing After Impacted Tooth Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Serap Keskin Tunc, Associate Professor Serap Keskin Tunc, Yuzuncu Yil University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: YYU-04/04.03.2020
Record Dates: First submitted 2023-09-14; First posted 2023-10-05 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Tooth Impaction; Tooth Diseases
Keywords: chlorhexidine, wisdom teeth, dental surgery
MeSH Terms: conditions — Tooth, Impacted; Tooth Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group using chlorhexidine toothpaste after wisdom tooth extraction (Experimental): 22 patients, 17 females and 5 males, 44 bilateral, similarly positioned fully impacted impacted lower third molars were extracted. Bilateral impacted wisdom teeth of the patients were randomly selected. After the operation, the experimental group received Dentasave 0.2% chlorhexidine toothpaste containing chlorhexidine
  Interventions: Procedure: Surgery of impacted mandibular wisdom teeth
- Control group using chlorhexidine-free toothpaste after wisdom tooth extraction (Placebo Comparator): Bilateral impacted wisdom teeth of the patients were randomly selected. After the operation, the control group was given toothpaste with the same ingredients as the study group but without chlorhexidine.
  Interventions: Procedure: Surgery of impacted mandibular wisdom teeth

INTERVENTIONS:
Procedure: Surgery of impacted mandibular wisdom teeth — All surgical procedures were performed by the same surgeon using the standard surgical technique described below. The anesthetic used was 4% articaine with 1:100,000 adrenaline. In all patients, a sulcus incision was made in the lower second molar and an envelope incision in the third molar region, the mucoperiosteal flap was removed, and extraction was performed with a bone elevator and a third molar elevator. If necessary, the impacted molar was incised with a high-speed dental handpiece and a fissure bur. The wound was irrigated with copious amounts of saline, and the wound edges were carefully sutured with simple 4.0 silk braided non-absorbable sutures.
  Other Names: Surgery of impacted mandibular wisdom teeth (the other side)

SUMMARY:
In this study, the postoperative clinical and microbiologic effects of chlorhexidine toothpaste and chlorhexidine-free toothpaste with the same content were compared after bilateral mandibular impacted third molar surgery. Similarly positioned fully impacted impacted lower third molars were extracted. Bilateral impacted wisdom teeth of the patients were randomly selected. After the operation, the experimental group received Dentasave 0.2% chlorhexidine toothpaste containing chlorhexidine and the control group received toothpaste with the same content but without chlorhexidine. Teeth were extracted by the same dentist at 14-day intervals. For microbiological analysis, saliva samples were taken before the first tooth extraction, before the second tooth extraction 14 days later and on the 28th day and sent to the microbiology laboratory. Wound healing, edema and trismus in both extractions were evaluated 1 week after tooth extraction. Wound healing was evaluated as good, acceptable and poor. VAS (Visual Analog Scale) was used for pain assessment and recorded 14 days after tooth extraction.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers with bilateral fully impacted mandibular wisdom teeth

Exclusion Criteria:

* Patients were excluded from the study if they did not understand the clinical procedures of the study,
* Had allergies or intolerance to any of the substances used in the study,
* Patients on anticoagulant or psychiatric treatment,
* Pregnant or breastfeeding,
* Patients using oral contraceptiveswere,
* Diabetic,
* Patients with periodontal disease or active infection
* Smokers of more than 10 cigarettes per day,
* Poor oral hygiene

Ages: 18 Years to 31 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Mouth opening measurements | 0-28 days
  the distance between the incisals of the patient's central teeth at maximal mouth opening.
Facial edema | 0-28 days
  Measurement between facial craniometric points (angulus-tragus, angulus-lateral canthus, angulus-nasal base, angulus-lateral canthus, and angulus-pogonion). The number of participants in the split mouth model was 22. A total of 44 impacted teeth were extracted and edema was measured before and 1 week after each extraction.
Wound healing | 0-28 days
  View of the wound site in the operation area. The REEDA scale was used for the clinical evaluation of the intraoral surgical field. This scale It includes five factors that indicate wound healing: Redness, Edema, Echymosis, Discharge, Approximation. Each of the recovery factors is evaluated by giving scores of 0, 1, 2 and 3 and the sum of the scores obtained as a result of the evaluation of these five categories constitutes the REEDA score. The lowest score is 0 and the highest score is 15.
Visual Analog Scale | 0-28 days
  A numerical rating scale VAS was used for pain analysis (0=no pain, 10=most severe pain). The pain levels at 24 hours, 48 hours and 1 week after the surgical procedure were recorded on the patient follow-up form by all patients who participated in the study by explaining that there was no pain at the "zero" level and the most severe pain known at the "10" level on the pain scale, which was organized as a 10 cm horizontal line on the prepared forms.
Microbiological analysis | 0-28 days
  Prior to extraction, a saliva sample was collected from the patient and placed in a sterile 1.5 ml Eppendorf tube and then stored in a -40 oC freezer. After surgical extraction, the patient was given toothpaste with the same content but without chlorhexidine. After a 14-day recovery period, the saliva sample was collected again without extracting the impacted tooth on the contralateral side, and tooth extraction was performed. After the second extraction, the patient was given Dentasave 0.2% Chlorhex toothpaste. The third saliva sample was collected on day 28 (14 days after the second tooth extraction).
  Saliva samples were stored in sterile universal containers (Eppendorf tubes) and sent to the microbiology laboratory less than 3 hours after collection on days 0, 14, and 28 of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yuzuncu Yil University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided